CLINICAL TRIAL: NCT03572595
Title: Diagnostic Accuracy of Positron Emission Tomography/ Computed Tomography With 18F-fluoro-2-deoxyglucose (18F- FDG PET/CT) in Patients With Colorectal Cancer
Brief Title: F-18 FDG- PETCT in Staging and Recurrent Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shymaa Mohamed, principle investigator, Assiut University
Other Study IDs: DPETCRC
Record Dates: First submitted 2018-06-09; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Colo-rectal Cancer; Recurrence
Keywords: FDG-PET/CT; Staging and restaging
MeSH Terms: conditions — Colonic Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Staging: Patients with pathologically proven colorectal cancer presented for pre-operative staging, underwent standard routine conventional radiological imaging i.e MRI , then will be subjected to be imaged by F-18 FDG-PET/CT from skullbase to midthigh, then interpretating the results of the hybrid PET/CT by two nuclear physicians then comparing with other conventional images.
  Interventions: Diagnostic Test: F-18 FDG-PET/CT
- Recurrent: Patients with treated colorectal cancer, suspecting of recurrence , will be subjected to be imaged by F-18 FDG-PET/CT from skull base to midthigh, interpretating the results of the hybrid PET/CT by two nuclear physicians.
  Then refer back to the treating physicians , another biopsy will be taken from the suspected recurrence and then results will be compared with hybrid PET/CT images.
  comparing the results with histopathology .
  Interventions: Diagnostic Test: F-18 FDG-PET/CT

INTERVENTIONS:
Diagnostic Test: F-18 FDG-PET/CT — imaging using Positron Emission Tomography/ Computed Tomography with 18F-fluoro-2-deoxyglucose (18F- FDG PET/CT) in Patients with colorectal cancer either for staging or suspecting recurrence

SUMMARY:
Colorectal cancer (CRC) is the fourth most frequently diagnosed cancer and the second leading cause of cancer death in the United States.

The overall relative 5-year survival is about 50%-60% but is highly dependent on disease stage at the time of diagnosis ranging from approximately 80% to only 3%.

Curative treatment comprises resection of the primary tumour combined with adjuvant chemotherapy in selected patients. In recent years there has been an increasing role for curative intended surgical or ablative intervention in limited metastatic disease, i.e., solitary or few metastases to the liver and/or the lungs. Accurate preoperative staging is of paramount importance for directing the most appropriate therapeutic options, for indicating prognosis and outcome, and to avoid futile operations.

DETAILED DESCRIPTION:
The use of imaging in the staging and restaging of colorectal cancers has been evolving and improving in the last two decades. Magnetic resonance imaging (MRI) is an accepted modality for staging of rectal cancer, allowing an accurate identification of transmural invasion of the mesorectal fat and mesorectal fascia involvement. Computed tomography (CT) significantly lacks resolution of soft tissue contrast so that its utility in T staging of rectal cancer is limited. Due to the higher sensitivity and specificity compared with CT,Positron Emission Tomography/ Computed Tomography with 18F-fluoro-2-deoxyglucose (FDG PET/CT) is recommended for use in a metastatic patients.

Pelvic MRI and 18F-FDG PET/CT are useful for staging and therapeutic management. Pelvic MRI allows for accurate definition of the distance to mesorectal fascia which is a predictor of the local recurrence rate, as well as for definition of the regional nodal status. 18F-FDG PET/CT also helps in evaluating the nodal status and is especially performed for the detection of distant metastases. MRI and 18F-FDG PET/CT are thus 2 complementary modalities for the initial staging of advanced rectal cancer.

Neoadjuvant therapies are performed for stage II and stage III rectal cancer. It has been shown that neoadjuvant therapy decreases local recurrence and increases survival. Therefore, correct preoperative staging has a critical role in determining whether patients should undergo neoadjuvant therapy.

The literature on the clinical use of FDG-PET/CT in colorectal cancer staging is fairly limited, but recent works have demonstrated some promise for optimizing the accuracy of initial staging by clarifying equivocal findings on conventional imaging in preoperative staging, and evaluating apparently limited metastatic disease before intervention .

It was reported that the use of FDG-PET/CT in this study changed the planned treatment strategy in a total of 30% of the patients. A change from palliative to curative or vice versa was seen in almost 10% of the patients.

PET/CT provides high accuracy for the detection and staging of liver lesions in CRC patients, PET led to a change in patient management in an average of 24 % of patients, including both exclusion from curative surgery and modification of the surgical approach.

Risk of local recurrence is substantial and correlates to the extension and grade of the tumor and to the nodal status at initial presentation. The guidelines also highlight the usefulness of PET/CT for restaging in the setting of a serially elevated carcinoembryonic antigen level (CEA), negative results on conventional imaging, and potentially resectable metachronous metastases documented by CT, MRI, or biopsy.It was reported that a high sensitivity and specificity of 18F-FDG PET/CT in detecting recurrent CRC, largely regardless of CEA levels, as well as they concluded that 18F-FDG PET/CT have high diagnostic value and can be used as the first choice in the detection of recurrent CRC in patients with unexplained rising CEA, even in patients with a recent normal routine CT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically proven colorectal cancer presented for pre-operative staging or restaging.
* Patients with treated colorectal cancer , suspecting recurrence .

Exclusion Criteria:

* Pregnancy.
* Patients with double primary.
* Expected life less than 3 months.
* Uncontrolled diabetes or elevated blood sugar more than 200 mg/dl.
* Severe medical condition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients daignosed with colorectal cancer , presented for pre-operative staging, so after doing the standard routine conevntional imaging , they will be sceduled to be imaged with F_18 FDG_PET/CT , hpothezied that the latter has potential promosing role in staging of those patients and lead to change of mangenent.
  As well, patients with treated colorectal cancer , under follow up, suspecting recurrence , will be sceduled to be iamged with F-18 FDG-PET/CT for determing is role in those patients.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
How many patients will be upstaged or downstaged by using pre-operative F-18 FDG_PET/CT in patients with colorectal cancer. | 2 weeks after the patients have been diagnosed and presented for treatment
  role of F-18 FDG_PET/CT in staging of colorectal cancer patient .

SECONDARY OUTCOMES:
Number of patients will be diagnosed recurrent colorectal cancer by using F-18 FDG_PET/CT in case of negative other conventional imaging. | one week
  which is better F-18 FDG_PET/CT or other conventional imaging

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Mekkay, PHD, Principal Investigator — Assiut University

REFERENCES:
- [Background] Chowdhury FU, Shah N, Scarsbrook AF, Bradley KM. [18F]FDG PET/CT imaging of colorectal cancer: a pictorial review. Postgrad Med J. 2010 Mar;86(1013):174-82. doi: 10.1136/pgmj.2009.079087. PMID 20237012
- [Background] Cerny M, Dunet V, Prior JO, Hahnloser D, Wagner AD, Meuli RA, Schmidt S. Initial Staging of Locally Advanced Rectal Cancer and Regional Lymph Nodes: Comparison of Diffusion-Weighted MRI With 18F-FDG-PET/CT. Clin Nucl Med. 2016 Apr;41(4):289-95. doi: 10.1097/RLU.0000000000001172. PMID 26828149
- [Background] Benson AB 3rd, Venook AP, Cederquist L, Chan E, Chen YJ, Cooper HS, Deming D, Engstrom PF, Enzinger PC, Fichera A, Grem JL, Grothey A, Hochster HS, Hoffe S, Hunt S, Kamel A, Kirilcuk N, Krishnamurthi S, Messersmith WA, Mulcahy MF, Murphy JD, Nurkin S, Saltz L, Sharma S, Shibata D, Skibber JM, Sofocleous CT, Stoffel EM, Stotsky-Himelfarb E, Willett CG, Wu CS, Gregory KM, Freedman-Cass D. Colon Cancer, Version 1.2017, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2017 Mar;15(3):370-398. doi: 10.6004/jnccn.2017.0036. PMID 28275037
- See also: Routine use of positron-emission tomography/computed tomography for staging of primary colorectal cancer: Does it affect clinical management? — https://doi.org/10.1186/1477-7819-11-49
- See also: Diagnostic value of 18F-FDG PET/CT as first choice in the detection of recurrent colorectal cancer due to rising CEA — https://doi.org/10.1186/s40644-015-0048-y